CLINICAL TRIAL: NCT01687322
Title: Long Term Follow-Up After Patients Underwent Total Hip Replacement
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, iri liebergall, Prof Meir (Iri) Liebergall, Chairman, Orthopedic Surgery Dept., Hadassah Medical Organization
Other Study IDs: lieb004-CTIL-HMO
Record Dates: First submitted 2012-08-23; First posted 2012-09-18 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Total Hip Replacement; Pain
Keywords: quality of life; functioning
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- total hip replacement, quality of life, functioning

SUMMARY:
The investigators want to contact patients that underwent total hip replacement for the past ten years. The investigators will ask them about their daily living, functioning and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. total hip replacement from 01.01.2002

Exclusion Criteria:

1. no

Ages: 28 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: men and women than underwent total hup replacment
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
quality of life | up to ten years
  quality of life will be assessed by the SF-12 questionnaire. We will compare between the results from the last visit to the current.

SECONDARY OUTCOMES:
functioning | up to ten years
  functioning will be assessed by the Harris Hip Score. We will compare between the results from the last visit to the current visit

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel